CLINICAL TRIAL: NCT02942979
Title: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking (MISSION) (QUE 15-284)
Brief Title: Maintaining Independence and Sobriety Through Systems Integration, Outreach, and Networking
Acronym: MISSION-HPACT
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: QUX 16-011; QUE 15-284 (Other: VAHSRD)
Record Dates: First submitted 2016-10-17; First posted 2016-10-24 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Co-Occurring Disorders; Homelessness; Substance Abuse Disorder; Mental Illness
Keywords: Facilitation; Implementation; Homelessness; Substance Use Disorder; Mental Illness; Co-Occurring Disorders; Veterans; Primary Care
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MISSION Implementation as Usual: Passive implementation or, IU for MISSION-Vet is comprised of a two-hour webinar training, along with key information on how to access and use the MISSION-Vet Treatment Manual and Consumer Workbook. The manual is posted on the web and available inside the VA on the National Center for Homelessness Among Veterans website or at missionmode.org. This passive implementation strategy has been used in previous studies
- Facilitation Implementation of MISSION: Facilitation is a comprehensive approach in which implementation experts partner with local staff to support implementation planning and to tailor adoption strategies to the local context. Facilitation gives attention to addressing individual- and organizational-level factors that can influence successful implementation of an evidence based practice with good fidelity.

SUMMARY:
This study seeks to implement wrap around services for Veterans suffering from co-occurring mental illness and substance use and who are homeless. It will compare Implementation as Usual of MISSION to Facilitation Implementation of MISSION.

DETAILED DESCRIPTION:
Background: Homeless Veterans often have multiple health care and psychosocial needs, including assistance with access to housing and health care, as well as support for ongoing treatment engagement. The Department of Veterans Affairs (VA) developed specialized Homeless Patient Alignment Care Teams (HPACT) with the goal of offering an integrated, "one-stop program" to address the Housing and Healthcare needs of Homeless Veterans. However, while 70% of HPACT's Veteran enrollees have co-occurring mental health and substance use disorders (COD), HPACT does not have a uniform, embedded treatment protocol for this subpopulation. One wraparound intervention designed to address the needs of homeless Veterans with COD which is suitable to be integrated into HPACT clinic sites is the evidence-based practice called Maintaining Independence and Sobriety through Systems Integration, Outreach, and Networking-Veterans Edition, or MISSION-Vet. Despite the promise of MISSION-Vet within HPACT clinics, implementation of an evidence based intervention within a busy program like HPACT can be difficult. The current study is being undertaken to identify an appropriate implementation strategy for MISSION-Vet within HPACT. The study will test the implementation platform called Facilitation and compared to implementation as usual (IU).

Aims: (1) Compare the extent to which IU or Facilitation strategies achieve fidelity to the MISSION-Vet intervention as delivered by HPACT homeless provider staff. (2) Compare the effects of Facilitation and IU strategies on the National HPACT Performance Measures. (3) Compare the effects of IU and Facilitation on the permanent housing status. (4) Identify and describe key stakeholders' (patients, providers, staff) experiences with, and perspectives on, the barriers to, and facilitators of implementing MISSION.

Design: Type III Hybrid modified stepped wedge implementation comparing IU to Facilitation across 7 HPACT teams in 3 sites in the greater Los Angeles VA system.

Discussion: Integrating MISSION-Vet within HPACT has the potential to improve the health of thousands of Veterans but, it is crucial to implement the intervention appropriately in order for it to succeed. The lessons learned in this protocol could assist with a larger roll-out of MISSION within HPACT.

ELIGIBILITY:
Inclusion Criteria:

* meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition diagnostic criteria of International Classification of Diseases, 10th Revision for a current substance abuse or dependence disorder, e.g.:

  * alcohol
  * marijuana
  * cocaine
* or poly substance use and a co-occurring mental illness that includes anxiety, mood, or a psychotic spectrum disorder
* is willing to participate in the service
* is empaneled in HPACT at one of the study sites

Exclusion Criteria:

* Does not meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Homeless Veterans in the Greater Los Angeles VA system
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Smelson, PsyD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Allen L. Gifford, MD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA; Sonya Emi Gabrielian, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yakovchenko V, McCullough MB, Smith JL, Gabrielian S, Byrne T, Bruzios KE, Koosis E, Smelson DA. Implementing a complex psychosocial intervention for unstably housed Veterans: A realist-informed evaluation case study. Implement Res Pract. 2021 Oct 26;2:26334895211049483. doi: 10.1177/26334895211049483. eCollection 2021 Jan-Dec. PMID 37090015
- [Derived] Smelson DA, Yakovchenko V, Byrne T, McCullough MB, Smith JL, Bruzios KE, Gabrielian S. Testing implementation facilitation for uptake of an evidence-based psychosocial intervention in VA homeless programs: A hybrid type III trial. PLoS One. 2022 Mar 17;17(3):e0265396. doi: 10.1371/journal.pone.0265396. eCollection 2022. PMID 35298514
- [Derived] Simmons MM, Gabrielian S, Byrne T, McCullough MB, Smith JL, Taylor TJ, O'Toole TP, Kane V, Yakovchenko V, McInnes DK, Smelson DA. A Hybrid III stepped wedge cluster randomized trial testing an implementation strategy to facilitate the use of an evidence-based practice in VA Homeless Primary Care Treatment Programs. Implement Sci. 2017 Apr 4;12(1):46. doi: 10.1186/s13012-017-0563-2. PMID 28376839
- See also: Describes the intervention. — http://www.missionmodel.org

RESULTS

PARTICIPANT FLOW:
Period: Step 0
Arm/Group | MISSION Implementation as Usual | Facilitation Implementation of MISSION
Started | 108 | 0
Completed | 108 | 0 (This is a stepped wedge design - all participants received both MISSION Implementation as Usual and Facilitation)
Not Completed | 0 | 0
Period: Step 1
Arm/Group | MISSION Implementation as Usual | Facilitation Implementation of MISSION
Started | 15 | 93
Completed | 15 | 93
Not Completed | 0 | 0
Period: Step 2
Arm/Group | MISSION Implementation as Usual | Facilitation Implementation of MISSION
Started | 0 | 108
Completed | 0 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants received both arms of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | MISSION Implementation as Usual | Facilitation Implementation of MISSION | Total
Number analyzed (Participants) | 108 | 0 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12) |  | 49 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only 77 of 108 responded to item
  Participants
    number analyzed (Participants) | 77 | 0 | 77
    Female | 37 |  | 37
    Male | 40 |  | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 0 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of MISSION Sessions Undertaken
Description: Number of MISSION Sessions delivered to Veterans
Time Frame: 12 months
Population: Stepped wedge design - all participants received both MISSION Implementation as Usual and Facilitation Implementation of MISSION
Measure: Number; unit: number of MISSION Sessions
Arm/Group | MISSION Implementation as Usual | Facilitation Implementation of MISSION
Number analyzed (Participants) | 108 | 108
number of MISSION Sessions | 0 | 574

ADVERSE EVENTS:
Time Frame: time of study entry until the end of study participation which was on average 1 year
Arm/Group | MISSION Implementation as Usual | Facilitation Implementation of MISSION
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/108
Other Adverse Events (participants affected / at risk) | 0/108 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02942979/Prot_SAP_000.pdf